CLINICAL TRIAL: NCT05697094
Title: Impact of Meditation on Improving Quality of Life Among Glaucoma Patients: An Electronic Pilot Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Monali Malvankar, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 119431
Record Dates: First submitted 2021-06-25; First posted 2023-01-25 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma; Depression; Anxiety; Sleep Disorder; Quality of Life
Keywords: Health-related quality of life; Glaucoma; Meditation
MeSH Terms: conditions — Glaucoma; Depression; Anxiety Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation to Remove Stress and Create A Proper System in Mind (Experimental): The study intervention will be administered to participants randomized to the intervention arm. The meditation intervention will be delivered virtually via the hospital-approved Microsoft Teams platform. Participants will be taught an evidence-based meditation technique which includes two online sessions (60 minutes/day) with a trained, experienced, and certified teacher of Prasanna Wellness, a non-profit service organization. Participants will learn how to respond to experiences that arise in meditation, will discuss what enhances or detracts from effective meditation, and review methods for meditating at home. The participants in the intervention arm will complete 60-minute follow-up sessions with the Prasanna Wellness staff which will include 33 minutes of guided meditation practice, and then a discussion of participants' experiences with meditation during the week, additional observations, and a review of relevant knowledge to support their home practice.
  Interventions: Behavioral: Meditation to Remove Stress and Create A Proper System in Mind
- Usual Care (No Intervention): Participants will continue with their usual care.

INTERVENTIONS:
Behavioral: Meditation to Remove Stress and Create A Proper System in Mind — Meditation to Remove Stress and Create A Proper System in Mind is a guided meditation.
  Other Names: Beyond Mindfulness Meditation
  Arms: Meditation to Remove Stress and Create A Proper System in Mind

SUMMARY:
Glaucoma is a chronic disease that causes loss of vision and potentially blindness as a result of optic nerve damage due to increased intraocular pressure. Currently, it is the leading cause of irreversible blindness worldwide1. In 2020, 4.1 million and 3.6 million adults over the age of 50 suffered from mild to severe visual impairment and blindness respectively induced by glaucoma1. However, these predictions are likely underestimated since glaucoma can remain asymptomatic until later stages in disease progression2.

There is a convincing body of evidence suggesting that there is a linear relationship between visual impairment and decreased quality of life (QOL) among glaucoma patients3. Furthermore, evidence from The National Health and Aging Trends Study suggests that this relationship may be bidirectional where older adults with visual impairment are more likely to suffer from mental illness and older adults with mental illness are more likely to suffer from visual impairment4. Mindfulness-based meditation is a promising non-pharmacological treatment that has been shown to reduce intraocular pressure and improve QOL in patients with glaucoma5.

A feasibility study will be conducted using a mixed-method design to assess the feasibility of delivering a meditation intervention online to enhance the QOL and mental health of glaucoma patients. Participants will be recruited and randomized in blocks of 10 and will undergo 1:1 randomization to the intervention arm or usual care arm. The purpose of this block randomization technique is to minimize the wait time between patient recruitment and study initiation. Participants in each arm will complete online questionnaires at patient recruitment, weeks 1, 3, 6, and 12 to measure self-reported health, depression symptoms, anxiety, and sleep quality using REDCap, an electronic data capturing system provided by Lawson Health Research Institute (LHRI).

ELIGIBILITY:
Inclusion Criteria

1. Patients diagnosed with mild glaucoma.
2. Patients aged 65-75.
3. Being able to provide valid informed consent to participate in the research study.
4. Being able to read and understand English.
5. Having no significant self-reported or physician-diagnosed mental health disorder.
6. Able to independently access a computer to participate in virtual meditation sessions.
7. Must be able to sit comfortably for 30-35 minutes without any major pain or discomfort, can hear well enough to follow verbal instructions when the eyes are closed, and be in good general physical health.

Exclusion Criteria

1. Inability to provide valid informed consent.
2. Significant communication barriers or lack of English proficiency that prevents participants from completing the questionnaires.
3. Severe depression as confirmed by a CES-D ≥ 24.
4. Having a lifetime diagnosis of self-reported other serious mental disorders, including bipolar I or II disorder, primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).
5. Self-reported substance abuse or dependence within the past 3 months.
6. Having acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months.
7. Having irreversible vision loss that prevents one from completing the questionnaires.
8. Participation in a study involving similar techniques.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The 12-item short form survey | Week 1, week 3, week 6, week 12
  The 12-Item Short Form Survey (SF-12) is a questionnaire that measures self-reported health. Scores are calculated by converting the sum of responses to a scale from 0 to 100 where a higher score indicates superior health. In addition, results can be summarised using the physical component summary (PCS) score and the mental component summary (MCS) score.

SECONDARY OUTCOMES:
Depression | Week 1, week 3, week 6, week 12
  Depression is a feeling of severe despondency and dejection. Depression will be measured using the Center for Epidemiological Studies - Depression (CES-D) score.
  The CES-D provides scores from 0 to 60. Higher scores indicate worse outcome.
Anxiety | Week 1, week 3, week 6, week 12
  Anxiety will be measured using Hospital Anxiety and Depression Scale - Anxiety (HADS-A) subscale.
  The HADS-A provides scores from 0-21. Higher scores indicate worse outcome.
Sleep quality | Week 1, week 3, week 6, week 12
  Sleep quality as measured using the Pittsburgh Sleep Quality Index (PSQI) scores. The PSQI provides scores from 0-21. Higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) collected in this study will not be available to other researchers (e.g., outside the primary research group). Since the primary research group has the necessary expertise to analyze the data and do not need any outside help.

REFERENCES:
- [Background] Atreya CE, Kubo A, Borno HT, Rosenthal B, Campanella M, Rettger JP, Joseph G, Allen IE, Venook AP, Altschuler A, Dhruva A. Being Present: A single-arm feasibility study of audio-based mindfulness meditation for colorectal cancer patients and caregivers. PLoS One. 2018 Jul 23;13(7):e0199423. doi: 10.1371/journal.pone.0199423. eCollection 2018. PMID 30036361
- [Background] Yunesian M, Aslani A, Vash JH, Yazdi AB. Effects of Transcendental Meditation on mental health: a before-after study. Clin Pract Epidemiol Ment Health. 2008 Nov 1;4:25. doi: 10.1186/1745-0179-4-25. PMID 18976496